CLINICAL TRIAL: NCT04337567
Title: A Prospective Randomized Trial for the Comparison of Procedural Characteristics and Long-term Effects of Radiofrequency Ablation and Balloon Cryoablation in Elderly Patients With Atrial Fibrillation
Brief Title: Radiofrequency Ablation Versus Balloon Cryoablation in Elderly Patients With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vivantes Netzwerk für Gesundheit GmbH (Other)
Responsible Party: Principal Investigator, Charalampos Kriatselis, Principal Investigator, Vivantes Netzwerk für Gesundheit GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS_RFCR_ELDPA_0120
Record Dates: First submitted 2020-03-08; First posted 2020-04-07 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation
Keywords: ablative treatment of atrial fibrillation; ballon cryoablation; radiofrequency ablation; elderly patients
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients over 75 years_RF ablation (Active Comparator): Patients randomized to receive pulmonary vein isolation by means of radiofrequency ablation.
  Interventions: Procedure: radiofrequency ablation
- Patients over 75 years_ballon cryoablation (Active Comparator): Patients randomized to receive pulmonary vein isolation by means of ballon cryoablation.
  Interventions: Procedure: ballon cryoablation

INTERVENTIONS:
Procedure: radiofrequency ablation — ablative treatment as allocated to radiofrequency ablation
  Arms: Patients over 75 years_RF ablation
Procedure: ballon cryoablation — ablative treatment as allocated to ballon cryoablation
  Arms: Patients over 75 years_ballon cryoablation

SUMMARY:
This study compares the procedural characteristics and effectivity of radiofrequency ablation and cryoablation in patients with atrial fibrillation that are 75 years or older.

DETAILED DESCRIPTION:
Radiofrequency and cryoballon ablation have been shown to be comparable to each other in terms of safety and effectivity in patients with atrial fibrillation. However, elderly patients have been underrepresented in the previous studies. The number of older patients with atrial fibrillation is high and the number of who undergo an ablation procedure for atrial fibrillation increases steadily. This prospective randomized trial compares the effectivity (recurrency of atrial arrhythmias) and periprocedural characteristics of the two established ablation methods in patients who are 75 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent symptomatic paroxysmal or persistent atrial fibrillation
* At the day of their inclusion in the study the patients have to have completed the 75th year of life

Exclusion Criteria:

* Dementia
* Presence of left atrial thrombus
* Left atrial volume> 50 ml/m²
* Renal failure (GFR≤ 30 ml/min)
* Comorbidity with an expected survival of 12 months or less.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
atrial arrhythmia recurrence | 1 year
  Number of Participants with recurrence of any atrial arrhythmia with a duration of 30 sec or longer 12 months after the ablative treatment

SECONDARY OUTCOMES:
procedural duration | periprocedural
  Duration of the whole procedure [min] inclusive preparation (from entrance to the EP lab till exit from the EP lab)
time to wake-up after propofol withdrawal | periprocedural
  Time from withdrawal of propofole till patient awake and fully oriented (time, place, person)
contrast medium dosis | periprocedural
  Amount of contrast medium used
Propofoldosis | periprocedural
  Propofoldosis needed for sedation
groin complications | up to 3 months after dismission from the hospital
  Number of Participants in each randomisation arm with groin complications (hematoma, av fistel, Aneuryma spurium, infection).
Neurological complications | 1 year
  Number of Participants in each randomisation arm with transient ischemic attack, cerebral insult, cerebral haemorrhage
vascular complications | 1 year
  Number of Participants in each randomisation arm with deep vein thrombosis, peripheral embolism.
duration of hospital staying [days] | 1 year
  duration of hospital staying: from admission till discharge in days

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Kriatselis, MD, Principal Investigator — Vivantes Clinic Neukölln
Locations (1):
- Vivantes Klinikum Neukölln, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No